CLINICAL TRIAL: NCT03518918
Title: Establishing the Diagnosis Standard and Analysis the Risk Factors of Premature Ovarian Insufficiency in Chinese Women： Multi-center, Prospective,Observational Study
Brief Title: Establishing the Diagnosis Standard and Analysis the Risk Factors of POI in Chinese Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Southern Medical University, China (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); Shenzhen Hospital of Southern Medical University (Other); Shen-Zhen City Maternity and Child Healthcare Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2016-141
Record Dates: First submitted 2017-06-13; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2017-05

CONDITIONS: Primary Ovarian Insufficiency
Keywords: Premature ovarian insufficiency; Diagnosis standard; Risk factors
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to establishing the diagnosis standard of POI and analyzing the risk factors in Chinese women.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. The POI guideline development group of ESHRE recommends the following diagnostic criteria: oligo/amenorrhea for at least 4 months and an elevated follicle stimulating hormone (FSH) level >25 mIU/mL on two occasion >4 weeks apart. But there still no diagnosis standard of POI in Chinese.The study aims to establishing the diagnosis standard of POI and analyzing the risk factors in Chinese women.

ELIGIBILITY:
Inclusion Criteria:

* Infertility
* The length of menstrual cycle longer than 35 days or shorter than/amenorrhea
* Serum FSH levels ≥10mIU/ml/ serum AMH levels ≤1.0pg/ml/ AFC ≤7, on at least two occasion >4 weeks apart

Exclusion Criteria:

* Polycystic Ovarian Syndrome
* other causes of amenorrhea

Ages: 12 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female under the condition of diminished ovarian reserve were enrolled in the study. The condition of diminished ovarian reserve may be the early stage of premature ovarian insufficiency.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of serum FSH levels | through study completion, an average of 3 months, assessed up to 48 months
  the serum FSH levels between day 2 to day 5 of menstrual cycle from date of recruit until the date of study completion or date of twice FSH level >25mIU/mL, whichever came first.
Menstruation situation | through study completion, an average of 3 months, assessed up to 48 months
  the length of the menstrual cycle from date of recruit until the date of study completion or date of twice FSH level >25mIU/mL, whichever came first.

SECONDARY OUTCOMES:
Change of Antral follicle count | through study completion, an average of 3 months, assessed up to 48 months
  the Antral follicle count between day 2 to day 5 of menstrual cycle from date of recruit until the date of study completion or date of twice FSH level >25mIU/mL, whichever came first.
Change of anti-mullerian hormone levels | through study completion, an average of 3 months, assessed up to 48 months
  the anti-mullerian hormone between day 2 to day 5 of menstrual cycle from date of recruit until the date of study completion or date of twice FSH level >25mIU/mL, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Shi-ling Chen, M.D, Ph.D, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Center for Reproductive Medicine, Department of Gynecology and Obstetrics, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China